CLINICAL TRIAL: NCT01065558
Title: A Safety and Pilot Activity Study of Ecopipam (PSYRX 101) in the Symptomatic Treatment of Self-Injurious Behavior in Subjects With Lesch-Nyhan Disease
Brief Title: Safety and Tolerability of the D1 Dopamine Receptor Antagonist Ecopipam in Patients With Lesch-Nyhan Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Psyadon Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Ecopipam and Lesch-Nyhan
Record Dates: First submitted 2010-02-06; First posted 2010-02-09 (Estimated); Results first posted 2013-04-18 (Estimated); Last update posted 2013-04-18 (Estimated); Status verified 2013-04

CONDITIONS: Lesch-Nyhan Disease
Keywords: Ecopipam; Lesch-Nyhan Disease; Safety; Self-Injurious Behavior
MeSH Terms: conditions — Lesch-Nyhan Syndrome; Self-Injurious Behavior | interventions — ecopipam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ecopipam 12.5 - 200 mg/day (Experimental): Patients were administered ecopipam on an escalated dosing schedule over 11 days starting at 12.5 mg/day and increasing to the maximal tolerated dose or to 200 mg/day.
  Interventions: Drug: Ecopipam

INTERVENTIONS:
Drug: Ecopipam — Tablets, once daily, for two weeks up to 200 mg/day
  Other Names: PSYRX101, SCH 39166

SUMMARY:
The purpose of this study is to determine the effects of ecopipam in patients with Lesch-Nyhan Disease (LND). Ecopipam specifically blocks the actions of one chemical in the brain that helps nerves talk to one another; ecopipam does this by stopping the chemical (dopamine) from binding to one of its family of receptors (i.e, the D1 family). LND is a very rare genetic disease. The sponsor is doing this study to find out what side effects ecopipam causes in LND patients, and whether ecopipam may be able to relieve the self-injurious behaviors seen in these patients.

ELIGIBILITY:
Inclusion Criteria

* Diagnosis of Lesch-Nyhan disease with moderate to severe Self- Injurious Behavior and are routinely restrained
* Male - 6 years of age and above
* Body weight greater than or equal to 44 pounds

Exclusion Criteria:

* Taking Neuroleptic or Dopamine Depleting medications
* Currently treated with medications for depression or seizures
* Impaired renal function
* Medical conditions that may interfere with completing the study

Ages: 6 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2010-02; Primary Completion 2011-01 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hyder A Jinnah, MD, Principal Investigator — Emory University; William L Nyhan, MD, Principal Investigator — University of California, San Diego
Locations (2):
- United States (2):
  - University of California at San Diego, San Diego, California
  - Emory Univesity, Atlanta, Georgia

REFERENCES:
- [Background] Chipkin RE, Iorio LC, Coffin VL, McQuade RD, Berger JG, Barnett A. Pharmacological profile of SCH39166: a dopamine D1 selective benzonaphthazepine with potential antipsychotic activity. J Pharmacol Exp Ther. 1988 Dec;247(3):1093-102. PMID 2905002

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited by the investigators according to the inclusion and exclusion criteria
Pre-assignment Details: No preassignment
Groups:
- Ecopipam (12.5- 200 mg/Day): Patients were given ecopipapm over an 11 day period as follows:
  day 1 12.5 mg/day day 2-3 25 mg/day day 4-5 50 mg/day day 6-9 100 mg/day day 9-11 200 mg/day
  Note: Doses were reduced as necessary to a previously tolerated dose if paitents reached doses that were not safely tolerable.
Period: Overall Study
Arm/Group | Ecopipam (12.5- 200 mg/Day)
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Lesch-Nyhan patients with moderate to severe self-injurious behaviors at the start of the study
Arm/Group | Ecopipam
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 4
  Between 18 and 65 years | 1
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 20.4 (17.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 5
Region of Enrollment [Number; unit: participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Clinically Significant Changes in Standard Laboratory Tests
Description: This study's primary outcome is the safety of ecopipam in Lesch-Nyhan patients as measured by standard clinical laboratory tests. The patients will also be observed and questioned about other side effects, such as whether they feel more or less tired.Standard clinical laboratory tests for liver, kidney and blood function were conducted. The normal ranges for each of these tests were different and are too numerous to be individually listed here. However, if any individual value were to be either three-times greater or lesser than the upper or the lower limit of the test, then that value was considered to have been changed.
Time Frame: Two weeks
Population: All patients were analyzed
Measure: Number; unit: Participants
Groups:
- Ecopipam Treated Patients: These were patients who had diagnoses Lesch-Nyhan Disease based either on their genetic changes or on changes of specific enzymes in their blood.
Arm/Group | Ecopipam Treated Patients
Number analyzed (Participants) | 5
Participants | 0

2. Secondary Outcome: Decrease in Self-injurious Behavior at End of Study (Two Weeks After Screening) Compared to Screening
Description: Change in the self-injurious subscale of the Behavior Problems Inventory (BPI). the BPI is a well-validate test to evaluate the frequency and severity of a patient's self-injurious behavior. Values range from 0 to 50, and a low score means few/less severe behaviors
Time Frame: Screening visit and end of study (two weeks)
Population: All patients who received any dose of ecopipam were in the analysis population
Measure: Mean (Standard Deviation); unit: Change in BPI score
Arm/Group | Ecopipam Treated Patients
Number analyzed (Participants) | 5
Change in BPI score | 22.5 (13.4)

ADVERSE EVENTS:
Time Frame: 12 days of active treatment and 28 days follow-up
Arm/Group | Ecopipam Treated Patients
Serious Adverse Events (participants affected / at risk) | 2/5
Other Adverse Events (participants affected / at risk) | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ecopipam Treated Patients (N=5)
Flank Pain (Renal and urinary disorders) | 1 (1) — Patient reported flank pain which was caused by a kidney stone. Investigator defined as not drug related, and resolved without incident. Patient received all doses and was not removed from study.
Respiratory Infection (Infections and infestations) | 1 (1) — Patient developed respiratory infection (pneumonia)following the trial. Investigator reported this as not related to ecopipam administration. Patient was briefly hosptialized and infection resolved.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ecopipam Treated Patients (N=5)
Sedation (Nervous system disorders) | 3 (3)
Dystonia (Nervous system disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 2 (2)

LIMITATIONS AND CAVEATS:
This was an open label trial of oral ecopipam in pediatric, adolescent and adult patients with Lesch-Nyhan Disease.In this population, ecopipam's safety and PK was similar to non-LND subjects.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less